CLINICAL TRIAL: NCT00128843
Title: Phase II Randomized, Multicenter, Crossover Clinical Trial for Administration of Exemestane vs. Anastrozole as First Line Treatment for Postmenopausal Patients With Hormone Receptor Positive Advanced Breast Cancer
Brief Title: Exemestane Versus Anastrozole as First Line Hormone Therapy in Postmenopausal Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2001-03
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; First line of hormone treatment; Postmenopausal women; Positive hormone receptor tumours
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exemestane (Experimental): 25mg/day per VO until progression disease, after this progression the patient could receive the another drug (comparator arm) ie Anastrozole by investigator decision
  Interventions: Drug: Anastrozole
- Anastrozole (Active Comparator): 1mg/day per VO until progression disease, after this progression the patient could receive the another drug (experimental arm) ie Exemestane by investigator decision
  Interventions: Drug: Exemestane

INTERVENTIONS:
Drug: Exemestane — 25mg/day until progression disease
  Other Names: Aromasil
  Arms: Anastrozole
Drug: Anastrozole — 1mg/day until progression disease
  Other Names: Arimidex
  Arms: Exemestane

SUMMARY:
This is a pivotal phase II, multicenter, open-label trial, designed to compare the efficacy of exemestane versus anastrozole as a first line treatment for advanced breast cancer. One hundred postmenopausal patients, with metastatic, positive hormone receptor breast cancer will be enrolled in this trial.

DETAILED DESCRIPTION:
The primary study endpoint is objective response rate. The study has been designed following Simon's test, with a p1-p0=0.15. p1 is the optimum level of activity of the experimental treatment (exemestane), and p0 is the minimum expected activity. In this study, p1 is 25% (25% of RR) and p0 is 10% (10% of RR). With an alpha error of 0.05 and a beta error of 0.1, Simon test establishes a first step of 21 patients per treatment arm. If at least 2 objective responses are observed in exemestane arm, recruitment will continue until 100 patients have been recruited. After this second recruitment phase, at least 7 objective responses must be observed to confirm the expected exemestane level of activity.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnoses of breast cancer.
* Postmenopausal women, defined as:

  * Bilateral surgical oophorectomy or amenorrhoea >= 5 years;
  * Age >= 56 years old and amenorrhoea >= 1 year;
  * Chemotherapy induced amenorrhoea >= 2 years;
  * Radiotherapy induced amenorrhoea at least 3 months before:
  * Age < 56 and < 5 years of amenorrhoea: follicle-stimulating hormone (FSH) levels to confirm postmenopausal status.
* Metastatic breast cancer (stage IV) or non-operable locally advanced breast cancer (stage IIIB).
* Positive estrogen and/or progesterone receptors as >10% cells or >10fmol/mg.
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Patients who have received adjuvant tamoxifen are eligible, if progression has been established at least 24 months since treatment start.
* Neoadjuvant chemotherapy is allowed if progression has been established at least 12 months after end of treatment.
* Patients may have received a first line of chemotherapy for advanced disease, but treatment must have ended at least 4 weeks before enrolment, and all acute toxicities must be resolved. Previous treatment with Herceptin is allowed.
* Normal haematological, hepatic and renal functions.
* Performance status ECOG of 0, 1, 2.
* Life expectancy superior to 3 months.
* Written informed consent.

Exclusion Criteria:

* Previous hormone treatment for metastatic disease.
* Previous treatment with aromatase inhibitors.
* Inflammatory breast cancer, or aggressive metastatic disease, or visceral lesions, or metastasis in the central nervous system (CNS).
* Non-measurable disease.
* Second malignancy except for basal skin carcinoma or cervical in situ carcinoma adequately treated. If other malignancies, patient must have a disease-free period superior to 5 years.
* Treatment with any investigational product in the 4 previous weeks.
* Patients with negative estrogen and progesterone receptor tumours.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2001-08 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) in both arms | up to 12 months
  Complete response plus partial response

SECONDARY OUTCOMES:
Time to progression | From date of randomization until the date of new documented progression, assessed up to 24 months
  Time from last patient included to progression disease
Time to progression after crossover | From date of crossover until the date of new documented progression, assessed up to 5 months
  Time from crossover (2nd line) to progression disease
Clinical benefit (1st line) | up to 6 months
  Completed response (CR) plus Partial Response (PR) plus Stable Diasease (SD) lasting ≥6 months
Clinical benefit after crossover (2nd line) | up to 6 months
  Completed response (CR) plus Partial Response (PR) plus Stable Diasease
Survival | up to 36 months
  Time from randomization of last patient included until death whatever cause.
Survival after crossover | up to 24 months
  Time from crossover until death whatever cause.
The Number of Participants Who Experienced Adverse Events (AE) | Until 30 days after the end of last patient study treatment (1st line)
  Patients who will receive at least one dose of Exemestane or Anastrozole will be evaluated for safety and toxicity. Safety will be assess by recording all clinical adverse events at each patient.
Toxicity after crossover | Until 30 days after the end of last patient study treatment (crossover: 2nd line)
  Patients who will receive at least one dose of Exemestane or Anastrozole will be evaluated for safety and toxicity. Safety will be assess by recording all clinical adverse events at each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Instituto Valenciano de Oncología
Locations (13):
- Spain (13):
  - Germans Trias i Pujol, Badalona, Barcelona
  - Clínico Universitario A Coruña (CHUAC), A Coruña, Galicia
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital Donostia, Donostia / San Sebastian, Guipúzcoa
  - H Comarcal de Barbastro, Barbastro, Huesca
  - H Puerto de Sagunto, Sagunto, Valencia
  - Hospital Clínico Universitario San Carlos, Madrid
  - Puerta de Hierro, Madrid
  - Ruber Internacional, Madrid
  - H Sant Camil, Tarragona
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Clínico Lozano Blesa, Zaragoza
  - H Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Llombart-Cussac A, Ruiz A, Anton A, Barnadas A, Antolin S, Ales-Martinez JE, Alvarez I, Andres R, Garcia Saenz JA, Lao J, Carrasco E, Camara C, Casas I, Martin M. Exemestane versus anastrozole as front-line endocrine therapy in postmenopausal patients with hormone receptor-positive, advanced breast cancer: final results from the Spanish Breast Cancer Group 2001-03 phase 2 randomized trial. Cancer. 2012 Jan 1;118(1):241-7. doi: 10.1002/cncr.26299. Epub 2011 Jun 29. PMID 21717449
- See also: Click here for more information about this study: GEICAM 2001-03 — http://www.geicam.org